CLINICAL TRIAL: NCT00238420
Title: A Phase I/II Trial of a Combination of Paclitaxel and Trastuzumab With Daily Irradiation or Paclitaxel Alone With Daily Irradiation Following Transurethral Surgery for Non-Cystectomy Candidates With Muscle-Invasive Bladder Cancer
Brief Title: Paclitaxel and Radiation Therapy With or Without Trastuzumab in Treating Patients Who Have Undergone Surgery for Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00730; NCI-2009-00730 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG-0524; CDR0000440988; RTOG 0524 (Other: Radiation Therapy Oncology Group); RTOG-0524 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-05

CONDITIONS: Bladder Urothelial Carcinoma; Stage I Bladder Cancer AJCC v6 and v7; Stage II Bladder Cancer AJCC v6 and v7; Stage III Bladder Cancer AJCC v6 and v7
MeSH Terms: interventions — Paclitaxel; Taxes; Radiotherapy; Radiation; Trastuzumab; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02

ARMS (2):
- Group I (paclitaxel, trastuzumab, radiation therapy) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, 15, 22, 29, 36, and 43 and trastuzumab IV over 90 minutes on day 1 and then over 30 minutes on days 8, 15, 22, 29, 36, and 43. Patients also undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, 43-47, and 50. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Radiation: Radiation Therapy; Biological: Trastuzumab
- Group II (paclitaxel, radiation therapy) (Experimental): Patients receive paclitaxel and undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, 43-47, and 50.
  Interventions: Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; Kanjinti; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera
  Arms: Group I (paclitaxel, trastuzumab, radiation therapy)

SUMMARY:
This phase I/II trial is studying the side effects of giving paclitaxel together with radiation therapy with or without trastuzumab and to see how well it works to kill any remaining tumor cells in patients who have undergone surgery for bladder cancer. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Paclitaxel may also make tumor cells more sensitive to radiation therapy. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving paclitaxel together with radiation therapy and trastuzumab may kill more tumor cells. Giving these treatments after surgery may kill any remaining tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the acute toxicity (=< 90 days from protocol treatment start) from chemoradiotherapy including paclitaxel +/- trastuzumab and irradiation in non-cystectomy patients with or without her2/neu overexpression.

SECONDARY OBJECTIVES:

I. To determine the ability of patients with bladder cancer who are non-cystectomy candidates to complete this treatment program.

II. To evaluate the efficacy of this treatment program in achieving a complete response of the primary tumor.

III. To measure the 5-year disease-free and overall survival of patients with bladder cancer treated with transurethral resection of the bladder followed by chemoradiotherapy.

IV. To estimate the value of tumor and/or serum biomarkers as predictors of initial tumor response and recurrence-free survival.

OUTLINE: This is a non-randomized, multicenter study. Patients are assigned to 1 of 2 treatment groups according to HER2/neu status (HER2/neu 2+ or 3+ staining [group 1] vs HER2/neu 0 or 1+ staining [group 2]).

GROUP I: Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, 15, 22, 29, 36, and 43 and trastuzumab (Herceptin®) IV over 90 minutes on day 1 and then over 30 minutes on days 8, 15, 22, 29, 36, and 43. Patients also undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, 43-47, and 50. Treatment continues in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive paclitaxel and undergo radiotherapy as in group 1.

After completion of study treatment, patients are followed at 4-5 weeks, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed primary transitional cell carcinoma (TCC) of the bladder

  * Histologic evidence of muscularis propria invasion
* Meets 1 of the following stage criteria:

  * Stage T2-4a; NX, N0, or N1; and M0 disease
  * Clinical stage T1, grade 3/3 disease AND requires definitive local therapy
* Tumor involvement of the prostatic urethra allowed provided the following criteria are met:

  * Tumor was visibly completely resected
  * No evidence of stromal invasion of the prostate
  * No evidence of distant metastases by chest x-ray (or chest CT scan) within 8 weeks prior to registration
  * No evidence of distant metastases by abdominal/pelvic CT scan (or MRI scan) within 8 weeks prior to registration
* Has undergone transurethral bladder resection (as thorough as is judged safely possible) within the past 3-8 weeks, including bimanual examination with tumor mapping
* Sufficient tumor tissue available for HER2/neu analysis
* Not a candidate for radical cystectomy
* Performance status - Zubrod 0-2
* Absolute neutrophil count >= 1,800/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 8.0 g/dL (transfusion or other intervention allowed)
* Bilirubin < 2.0 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) < 2.5 times upper limit of normal
* No hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* Creatinine =< 3.0 mg/dL
* Left ventricular ejection fraction (LVEF) >= 40% by multigated acquisition scan (MUGA) scan or echocardiogram
* No unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
* No transmural myocardial infarction within the past 6 months
* Not pregnant or nursing
* No nursing for 6 months after completion of study treatment (for patients receiving trastuzumab [Herceptin®])
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* Able to tolerate systemic chemotherapy and pelvic radiotherapy
* No other invasive malignancy within the past 3 years except nonmelanoma skin cancer
* No history of allergic reaction to study drugs
* No history of inflammatory bowel disease
* No acute bacterial or fungal infection requiring IV antibiotics
* No AIDS
* No other severe active comorbidity
* No prior systemic chemotherapy with anthracyclines or taxanes
* No prior systemic chemotherapy for TCC
* No prior pelvic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-07-26 (Actual); Primary Completion 2014-02-05 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. D Michaelson, Principal Investigator — Radiation Therapy Oncology Group
Locations (184):
- United States (180):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - The Reverend Roger Patrick Dorcy Cancer Center at Saint Mary-Corwin Medical Center, Pueblo, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Saint Francis Hospital - Wilmington, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Singing River Hospital, Pascagoula, Mississippi
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Institute-Summerlin Campus, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Saint Francis Hospital, Federal Way, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - London Regional Cancer Program, London, Ontario
  - McGill University Department of Oncology, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After patient registration, sites submitted tissue to central her2/neu evaluation. If tissue was evaluable and a patient continued on study, then treatment arm was assigned. Seventy-six patients were registered and 6 did not continue to treatment assignment: 2 patient withdrawal, 2 protocol violation, 1 progressive disease, 1 institutional error.
Groups:
- HER2+ :RT, Paclitaxel, and Trastuzumab: Paclitaxel and trastuzumab chemotherapy with concurrent with radiation therapy
- HER2- :RT and Paclitaxel: Paclitaxel chemotherapy concurrent with radiation therapy
Period: Overall Study
Arm/Group | HER2+ :RT, Paclitaxel, and Trastuzumab | HER2- :RT and Paclitaxel
Started | 22 | 48
Completed | 21 (Subjects with data available for the primary analysis are considered to have completed the study.) | 47 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who started protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | HER2+ :RT, Paclitaxel, and Trastuzumab | HER2- :RT and Paclitaxel | Total
Number analyzed (Participants) | 21 | 47 | 68
Age, Continuous [Median (Full Range); unit: years] | 80 [51 to 86] | 73 [53 to 90] | 75 [51 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 19 | 36 | 55

OUTCOME MEASURES:

1. Primary Outcome: Acute Treatment-related Toxicity
Description: In each group, the number of patients was tabulated by type and grade (gr) of treatment-related toxicity (CTCAE v3.0). Only the following types of toxicity within 90 days of treatment start were considered: ≥ gr4 neutropenia, ≥ gr4 febrile neutropenia, ≥ gr3 diarrhea, ≥ gr3 nausea/vomiting, ≥ gr3 thrombocytopenia, ≥ gr3 renal, pulmonary, hepatic, or neurologic toxicity, ≥ gr3 rectal or genitourinary bleeding, ≥ gr3 left ventricular failure, or ≥ gr2 other cardiac toxicity. The study was designed to estimate the rate of acute treatment-related toxicity separately in each group of patients. Using the Fleming's one-sample multiple test procedure with Type I and II errors each set at 10%, 40 cases/group were required to reject the null hypothesis that the true toxicity rate is greater than 25% in favor of the alternative hypothesis that the true rate is no more than 10%. Six or more patients with the designated toxicities out of 40 would result in rejecting the null hypothesis.
Time Frame: From start of protocol treatment to 90 days
Population: All eligible patients who started study treatment
Measure: Number; unit: participants
Arm/Group | HER2+ :RT, Paclitaxel, and Trastuzumab | HER2- :RT and Paclitaxel
Number analyzed (Participants) | 21 | 47
participants | 7 | 14

2. Secondary Outcome: Treatment Completion
Description: The number of patients within each group who completed all elements of protocol treatment are reported.
Time Frame: From registration to end of treatment; up to 64 days."
Population: All eligible patients who started study treatment
Measure: Number; unit: participants
Arm/Group | HER2+ :RT, Paclitaxel, and Trastuzumab | HER2- :RT and Paclitaxel
Number analyzed (Participants) | 21 | 47
participants | 13 | 34

3. Secondary Outcome: Complete Response to Treatment
Description: The number of patients within each group who achieved a complete response to protocol treatment by 12 weeks are reported. Complete response is defined as no gross tumor at cystoscopy or negative biopsies or both by week 12 after completion of protocol treatment.
Time Frame: At 12 weeks from treatment start
Population: All eligible patients who started treatment and had an evaluation to assess response by 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2+ :RT, Paclitaxel, and Trastuzumab | HER2- :RT and Paclitaxel
Number analyzed (Participants) | 13 | 33
percentage of participants | 61.5 [31.6 to 86.1] | 57.6 [39.2 to 74.5]

4. Secondary Outcome: Progression-free Survival
Description: Disease (failure) is defined as any bladder cancer progression determined by all measures of disease including physical exam, imaging, and biopsies. Disease-free survival time is defined as time from treatment start to the date of first progression, death, or last known follow-up (censored). Disease-free survival rates are estimated using the Kaplan-Meier method. Analysis occurred after all patients had been on study for at least 5 years. This is a non-randomized phase I/II trial in which the two patient groups are not compared.
Time Frame: From start of treatment to last follow-up. Maximum follow-up at time of analysis was 9.9 years.
Population: Eligible participants who started treatment. (This population changed since the initial analysis: 3 participants first thought to be eligible were later determined to be ineligible.)
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | HER2+ :RT, Paclitaxel, and Trastuzumab | HER2- :RT and Paclitaxel
Number analyzed (Participants) | 20 | 45
years | 1.1 [0.6 to 2.8] | 0.8 [0.4 to 3.0]

5. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as time from treatment start to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated using the Kaplan-Meier method. Analysis occurred after all patients had been on study for at least 5 years. This is a non-randomized phase I/II trial in which the two patient groups are not compared.
Time Frame: From the date of treatment started to death, assessed up to at least 5 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | HER2+ :RT, Paclitaxel, and Trastuzumab | HER2- :RT and Paclitaxel
Number analyzed (Participants) | 20 | 45
years | 2.8 [1.1 to 4.4] | 2.0 [1.1 to 8.5]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events.
Arm/Group | HER2+ :RT, Paclitaxel, and Trastuzumab | HER2- :RT and Paclitaxel
Serious Adverse Events (participants affected / at risk) | 6/21 | 15/47
Other Adverse Events (participants affected / at risk) | 20/21 | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HER2+ :RT, Paclitaxel, and Trastuzumab (N=21) | HER2- :RT and Paclitaxel (N=47)
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Myocardial ischemia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Supraventricular arrhythmia NOS (Cardiac disorders) | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Diarrhea NOS (Gastrointestinal disorders) | 4 | 3
Enteritis (Gastrointestinal disorders) | 0 | 1
Proctitis NOS (Gastrointestinal disorders) | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 0 | 1
Edema: limb (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Sudden death (General disorders) | 0 | 1
Hepatobiliary/pancreas - Other (Hepatobiliary disorders) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Urinary tract NOS (Infections and infestations) | 0 | 1
Kidney infection NOS (Infections and infestations) | 0 | 1
Pneumonia NOS (Infections and infestations) | 0 | 1
Urinary tract infection NOS (Infections and infestations) | 1 | 2
Vascular access NOS complication (Injury, poisoning and procedural complications) | 0 | 2
Leukopenia NOS (Investigations) | 0 | 1
Lymphopenia (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Personality change (Psychiatric disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urethral pain (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hematoma (Vascular disorders) | 1 | 0
Hypotension NOS (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HER2+ :RT, Paclitaxel, and Trastuzumab (N=21) | HER2- :RT and Paclitaxel (N=47)
Blood/bone marrow - Other (Blood and lymphatic system disorders) | 3 | 3
Hemoglobin (Blood and lymphatic system disorders) | 15 | 25
Atrial fibrillation (Cardiac disorders) | 2 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 2 | 7
Constipation (Gastrointestinal disorders) | 4 | 12
Diarrhea NOS (Gastrointestinal disorders) | 12 | 37
Flatulence (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 5 | 16
Proctitis NOS (Gastrointestinal disorders) | 3 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 3
Vomiting NOS (Gastrointestinal disorders) | 4 | 10
Edema: limb (General disorders) | 4 | 12
Fatigue (General disorders) | 15 | 39
Pain - Other (General disorders) | 2 | 2
Pyrexia (General disorders) | 0 | 4
Infection with unknown ANC: Urinary tract NOS (Infections and infestations) | 2 | 1
Opportunisitic infection (Infections and infestations) | 2 | 1
Urinary tract infection NOS (Infections and infestations) | 1 | 6
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 1 | 7
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 2
Blood bilirubin increased (Investigations) | 2 | 2
Blood creatinine increased (Investigations) | 6 | 13
Leukopenia NOS (Investigations) | 10 | 15
Lymphopenia (Investigations) | 8 | 10
Metabolic/laboratory - Other (Investigations) | 3 | 1
Neutrophil count (Investigations) | 5 | 4
Platelet count decreased (Investigations) | 5 | 10
Prothrombin time prolonged (Investigations) | 2 | 2
Weight decreased (Investigations) | 4 | 12
Anorexia (Metabolism and nutrition disorders) | 8 | 14
Dehydration (Metabolism and nutrition disorders) | 4 | 5
Hyperglycemia NOS (Metabolism and nutrition disorders) | 6 | 11
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 10
Hypokalemia (Metabolism and nutrition disorders) | 1 | 7
Hyponatremia (Metabolism and nutrition disorders) | 4 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 6
Dysgeusia (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 0 | 3
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 8
Anxiety (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 4 | 1
Bladder pain (Renal and urinary disorders) | 3 | 9
Bladder spasm (Renal and urinary disorders) | 1 | 6
Bladder stenosis (Renal and urinary disorders) | 2 | 0
Cystitis NOS (Renal and urinary disorders) | 12 | 17
Pollakiuria (Renal and urinary disorders) | 12 | 24
Proteinuria (Renal and urinary disorders) | 2 | 0
Renal/genitourinary - Other (Renal and urinary disorders) | 3 | 2
Ureteric obstruction (Renal and urinary disorders) | 1 | 4
Urethral pain (Renal and urinary disorders) | 0 | 4
Urinary bladder hemorrhage (Renal and urinary disorders) | 4 | 9
Urinary incontinence (Renal and urinary disorders) | 3 | 6
Urinary retention (Renal and urinary disorders) | 2 | 4
Pelvic pain NOS (Reproductive system and breast disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rhinitis allergic NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 7
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 1 | 4
Hypertension NOS (Vascular disorders) | 2 | 1
Hypotension NOS (Vascular disorders) | 2 | 5

LIMITATIONS AND CAVEATS:
Accrual of patients with her2/neu overexpression stopped early due to unmet targeted accrual goals, with 22 subject accrued out of 40 planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less